

## Protocol Synopsis

| <b>7</b> 1 | |
|---|---|
| Study Title | A multi-center, open, longitudinal, observational study to assess the treatment trend and the |
| | proportion of target blood pressure attainment in patients whose antihypertensive regimens are |
| | changed to angiotensin II receptor blocker-based therapy |
| | Study Short Title: FRESH study FimasaRtan-basEd BP Targets after Drug SwitcHing |
| Sponsor | Boryung Pharmaceutical Co., Ltd. |
| Study Objectives | The recent hypertension clinical practice guidelines published by American College of |
| | Cardiology (ACC) and American Heart Association (AHA) reduced the target BP to 130/80 |
| | mmHg, indicating the needs for more aggressive efforts in hypertension treatment. However, |
| | studies in Koreans must be preceded before applying such new overseas guidelines; thus, this |
| | study has been designed to establish clinical materials reflecting treatment setting in Korea. In |
| | this study, patients with uncontrolled hypertension whose antihypertensive regimens are changed |
| | to ARB-based therapy (ARB monotherapy or ARB-containing combination therapy) will be |
| | followed to assess the treatment trend, treatment effect, and risk of cardiovascular disease. |
| Sample Size | Approximately 5,000 subjects |
| Subject | ① Provided written consent to the use of personal information after receiving the explanation |
| Inclusion Criteria | of the objective, methodology, etc. of this clinical study |
| | ② Male or female adults ≥ 19 years who are diagnosed with essential hypertension |
| | 3 Receiving outpatient treatment at the time of study enrollment |
| | ④ Patients with hypertension uncontrolled by existing antihypertensive drugs (including ARB) |
| | whose antihypertensive regimens decided and scheduled to be changed to ARB |
| | monotherapy or ARB-containing combination therapy (the result of the arm with a higher |
| | mean BP [systolic BP preferred] when measured twice with at least a 2-minute interval in |
| | both arms at the medical office on the study enrollment date, will become the reference) |
| | ➤ Definition of uncontrolled hypertension: Target BP (SBP <140 mmHg and DBP <90 |
| | mmHg) not achieved even after the treatment using the existing antihypertensive drugs |
| | for 4 weeks or longer |
| Subject | ① Patients who were hospitalized or are scheduled to be hospitalized 4 weeks before or after |
| Exclusion Criteria | the study enrollment date |
| | ② Patients with suspected or confirmed secondary hypertension |
| | ③ Pregnant or breast-feeding women |
| | ④ Patients who received investigational product within 12 weeks or are scheduled to |
| | participate in another clinical study while participating in this study |
| | ⑤ Patients who are determined inappropriate for participating in the study by investigators for |
| | other reasons |
| Statistical Analysis | Analysis of Primary Endpoints |
| Methods | Frequency and proportion of patients who attain the target BP at Week 12 after the |
| | treatment regimen change will be calculated and the 95% confidence interval for the |

Protocol No.: BR-FMS-OS-404 Version 1.2, 2018.12.18



proportion will be provided.

## Analysis of Safety Data

- Incidence and characteristics of antihypertensive drug related adverse drug reactions
  For adverse drug reactions (ADRs) related to antihypertensive drugs, the number of subjects, incidence, 95% confidence interval for the incidence, and number of cases will be provided.
- Serious adverse events/adverse drug reactions
  For serious adverse events and serious adverse drug reactions, the number of subjects, incidence, 95% confidence interval for the incidence, and number of cases will be provided.